CLINICAL TRIAL: NCT00238485
Title: A 52-week, Open Label Extension Study to Evaluate the Safety and Tolerability of Licarbazepine 750 - 2000 mg/d in the Treatment of Manic Episodes of Bipolar I Disorder.
Brief Title: An Open-label Extension Study to Evaluate the Safety and Tolerability of Licarbazepine 750-2000 mg/d in the Treatment of Manic Episodes of Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLIC477D2302E1
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder
MeSH Terms: interventions — 10,11-dihydro-10-hydroxy-5H-dibenz(b,f)azepine-5-carboxamide

INTERVENTIONS:
Drug: Licarbazepine

SUMMARY:
This extension study is designed to investigate the long-term safety and tolerability of licarbazepine 750-2000 mg/d over 52 weeks in patients who completed the 6-week double-blind study CLIC477D2302.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent provided prior to participation in the extension study.
* successful completion of the study CLIC477D2302
* willingness and ability to comply with all study requirements

Exclusion Criteria:

* premature discontinuation from the study CLIC477D2302
* failure to comply with the study CLIC477D2302 protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of licarbazepine with respect to adverse events, serious adverse events, changes in laboratory values, ECGs and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Care information, Study Chair — 862-778-8300